CLINICAL TRIAL: NCT06006364
Title: Investigation of the Effect of Nomophobia on Musculoskeletal System and Sleep
Status: Completed | Type: Observational
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Other Study IDs: Uskudar55
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Dependence
Keywords: nomophobia; sleep
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1.Group: Nomophobia Level:none
  Interventions: Other: Survey
- 2.Group: Nomophobia Level: mild
  Interventions: Other: Survey
- 3.Group: Nomophobia Level: medium
  Interventions: Other: Survey
- 4.Group: Nomophobia Level: extreme
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — The scales and forms used are respectively:
  1. Demographic Information Form
  2. Nomophobia Scale
  3. Cornell Musculoskeletal Disorder Questionnaire
  4. Smart phone Addiction Scale
  5. Pittsburgh Sleep Quality Index
  6. International Physical Activity Survey
  7. McGill Melzack Pain Questionnaire

SUMMARY:
The aim of this study; Investigation of the effects on the musculoskeletal system and sleep by determining the nomophobia levels of individuals between the ages of 18-25.

DETAILED DESCRIPTION:
The research was planned as a quantitative research. Data collection was done online.

The scales and forms used are as follows:

1. Demographic Information Form
2. Nomophobia Scale
3. Cornell Musculoskeletal Disorder Questionnaire
4. Smart phone Addiction Scale
5. Pittsburgh Sleep Quality Index
6. International Physical Activity Survey
7. McGill Melzack Pain Questionnaire

Questionnaires will be sent to the participants online by invitation. Participants will be asked to participate in the study by reaching them through social media, mail or mobile phone applications. The data obtained will be analyzed statistically.

ELIGIBILITY:
Inclusion Criteria:

* To have accepted the voluntary consent form that requires participation in the survey study.
* Being a smart phone user

Exclusion Criteria:

* Not accepting the volunteer consent form
* Having undergone previous surgery
* Being on antidepressants.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: people with whom we were able to create the survey and who met the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
Nomophobia Scale | 2 days
  The Nomophobia Scale was itemized according to a 7-point Likert type. Out of 20 items in total consists of. The scale has four sub-dimensions: Lack of Access to Information (4 items), Losing Connection (5 items), Inability to Communicate (6 items), and Comfort Inability to feel (5 items).
Cornell Musculoskeletal Disorder Questionnaire | 2 days
  The questionnaire was conducted in 11 body regions (neck, right and left shoulder, upper arm, forearm and wrist, back and waist region) includes questions about the frequency of musculoskeletal disorders (pain/pain/discomfort), the severity of these disorders, and whether they interfere with work.
Smart phone Addiction Scale | 2 days
  It is a scale developed to measure the risk of smart phone addiction, consisting of 10 items and evaluated with a six-point Likert scale. Scale items were scored from 1 to 6. Scale scores range from 10 to 60. As the score obtained from the test increases, it is considered that the risk for addiction increases.
Pittsburgh Sleep Quality Index | 2 days
  It is a 19-item self-report scale that evaluates sleep quality and impairment over the past month. It consists of 24 questions, 19 questions are self-report questions, 5 questions are questions to be answered by the spouse or roommate. The 18 scored questions of the scale consist of 7 components. Subjective Sleep Quality, Sleep Latency, Sleep Duration, Habitual Sleep Efficiency, Sleep Disorder, Sleeping Drug Use and Daytime Dysfunction. Each component is evaluated over 0-3 points. The total score of the 7 components gives the scale total score. The total score ranges from 0 to 21. A total score greater than 5 indicates "poor sleep quality".
International Physical Activity Questionnaire Short Form | 2 days
  The questionnaire consisting of seven questions including the activities of the last seven days was prepared by the individuals themselves.
  self-applicable and provides information about the time people spend in moderate to vigorous activities
McGill Melzack Pain Questionnaire | 2 days
  Pain Questionnaire consists of four parts. With the McGill Melzack Pain Questionnaire, the location of the pain, the feeling it creates in the individual, its relationship with time, its severity and the level of livable pain for the individual are determined.

CONTACTS AND LOCATIONS:
Overall Officials: Melek ÖZCAN, Study Chair — Uskudar University
Locations (1):
- Uskudar Üniversity, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhattacharya S, Bashar MA, Srivastava A, Singh A. NOMOPHOBIA: NO MObile PHone PhoBIA. J Family Med Prim Care. 2019 Apr;8(4):1297-1300. doi: 10.4103/jfmpc.jfmpc_71_19. PMID 31143710
- [Background] Kuscu TD, Gumustas F, Rodopman Arman A, Goksu M. The relationship between nomophobia and psychiatric symptoms in adolescents. Int J Psychiatry Clin Pract. 2021 Mar;25(1):56-61. doi: 10.1080/13651501.2020.1819334. Epub 2020 Sep 17. PMID 32940094
- [Background] Notara V, Vagka E, Gnardellis C, Lagiou A. The Emerging Phenomenon of Nomophobia in Young Adults: A Systematic Review Study. Addict Health. 2021 Apr;13(2):120-136. doi: 10.22122/ahj.v13i2.309. PMID 34703533
- [Background] Rahme C, Hallit R, Akel M, Chalhoub C, Hachem M, Hallit S, Obeid S. Nomophobia and temperaments in Lebanon: Results of a national study. Perspect Psychiatr Care. 2022 Oct;58(4):1607-1612. doi: 10.1111/ppc.12968. Epub 2021 Nov 6. PMID 34741546
- [Background] Jahrami HA, Fekih-Romdhane F, Saif ZQ, Alhaj OA, AlRasheed MM, Pandi-Perumal SR, BaHammam AS, Vitiello MV. Sleep dissatisfaction is a potential marker for nomophobia in adults. Sleep Med. 2022 Oct;98:152-157. doi: 10.1016/j.sleep.2022.07.001. Epub 2022 Jul 11. PMID 35868112